CLINICAL TRIAL: NCT02957240
Title: Graded Motor Imagery for Women at Risk for Developing Type I CRPS Following Closed Treatment of Distal Radius Fractures: A Pilot Randomized Comparative Effectiveness Trial
Brief Title: Graded Motor Imagery for Women at Risk for Developing Type I CRPS Following Closed Treatment of Distal Radius Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: American Hand Therapy Foundation (Unknown); Fairview Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OT-2016-24458
Record Dates: First submitted 2016-10-25; First posted 2016-11-07 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Musculoskeletal Pain; Fractures, Closed; Distal Radius Fracture; Complex Regional Pain Syndromes
Keywords: Forearm [A01.378.800.585]; Radius [A02.835.232.087.090.700]; Motor Skills [F02.808.260]; Task Performance and Analysis [F02.808.600]; Casts, Surgical [E07.858.442.660.430.500]; Splints [E07.858.690.725.430.750]; motor representation techniques; mirror therapy; Women [M01.975]
MeSH Terms: conditions — Musculoskeletal Pain; Fractures, Closed; Wrist Fractures; Complex Regional Pain Syndromes | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Active Comparator): Four clinic-based intervention sessions where the focus will be on home program competency and advancement and standard home program 3x daily for 15 minutes.
  Interventions: Behavioral: Standard Care
- Standard Care and Motor Representation Techniques (Experimental): 4 clinic-based intervention sessions including 'standard care' intervention in addition to a 'movement representation' intervention. Home Program for Standard Care and Motor Representation 3x daily for 30 minutes.
  Interventions: Behavioral: Standard Care; Behavioral: Motor Representation Techniques

INTERVENTIONS:
Behavioral: Standard Care — This group will partake in 4 clinic-based intervention sessions (one 1-hr. and 3 subsequent 30-minute sessions) where the focus will be on home program competency/advancement. Session 1 will occur within 1 week of cast treatment, session 2 in week 2, session 3 in week 4, and session 4 in week 5.
  Home program (3x daily, 15 minutes) to include 10 repetitions of active thumb opposition, active thumb radial abduction, intrinsic minus active stretches, flat fist and composite, finger extension, Elbow flexion and extension, Shoulder scapular rolls, and glenohumeral circumduction.
  Edema will be addressed through strict elevation when at rest and every 10 minutes on the hour. When resting in a seated or supine position, clients will be instructed to use pillows to accomplish elevation and to keep elbows in an extended position. Instructions for elevation will be provided immediately following orthopaedic intervention. Strict elevation will be recommended for the first 72 hours of the injury.
Behavioral: Motor Representation Techniques — Those in this group will receive 4 clinic-based intervention session (one 1-hr. and three subsequent 30-minute sessions) where the focus will be on home program competency and advancement. Session 1 will occur within 1 week of cast treatment, session 2 in week 2, session 3 in week 4, and session 4 in week 5.
  Home Program will be performed 3x daily for 15 minutes. A Motor Representation Technique (i.e., modified GMI) protocol described by Lagueux et al. will be employed. As originally designed the program was broken into three stages 1) Laterality, 2) Explicit Motor Imagery, 3) Mirror therapy with unaffected hand only and 4) Mirror Therapy with bilateral hands. For the purpose of this study, and given the restraint offered by cast immobilization, the 4th phase will not be used. Each phase will require 1-2 weeks and will be progressed at the discretion of the hand therapist interventionist.
  Arms: Standard Care and Motor Representation Techniques

SUMMARY:
Nearly 2 out of 10 women will sustain a distal forearm fracture throughout their lifespan.Recent longitudinal studies illustrate that as many as 1/3 of all persons who undergo closed reduction and casting for distal radius fractures (DRF) go on to develop type 1 complex regional pain syndrome (CRPS). Graded motor imagery (i.e., motor imagery and mirror therapy), a movement representation technique, is strongly supported in the literature as a treatment of CRPS and has recently been suggested as a potential strategy to prevent its onset. Other complications include disability, wrist/forearm tightness and sensorimotor changes.

The investigators propose that an early intervention protocol which includes graded motor imagery (GMI) will improve the pain, functional and upper limb sensorimotor outcomes of persons following closed reduction and casting of DRF relative to a standard of care intervention.

DETAILED DESCRIPTION:
Distal radius fractures (DRF) account for nearly one-fifth of all fractures in older adults with women sustaining them at a rate of 5 to 1 relative to their male counterparts. The majority of DRF occur as a result of low impact injuries to the wrist with the hand being outstretched and are most often managed via closed treatment and cast immobilization The aftereffects of these injuries include pain, distal upper limb immobility, distal sensorimotor changes, hand weakness, edema, and type I complex CRPS development. Women, those sustaining low-force injuries, and those who undergo closed treatment and cast immobilization of the DRF, are at increased risk for developing type I CRPS. Given that alterations in the brain's somatosensory strip likely influence CRPS development, a newer intervention, graded motor imagery, is being used to restore the affected limbs cortical representation to its typical state. Beyond pain reduction, the implications of this type of approach also include restoring sensorimotor function to the affected limb. Evidence supports that these interventions can impact CRPS symptoms as well as motor function but only after they've developed. To date, there is no literature exploring how these techniques, specifically graded motor imagery, can be applied to prevent or mitigate the aforementioned aftereffects of DRF in women.

To this end the investigators propose to pilot a 6-week randomized comparative effectiveness trial, where the modified graded motor imagery program + standard of care group is compared to a standard of care (SOC) control group. Immediately following cast immobilization, the intervention group and control group will each participate in one 1-hr and three 30-minute clinic-based sessions and 15 minute home programs three times daily. Blinded assessments will occur at baseline, 3 weeks, cast removal, and one and 3 months after cast removal and will include pain, sensorimotor, edema, and CRPS diagnostic outcomes.

The project's aims are to: 1) determine the feasibility of recruiting, enrolling, treating, and following participants and 2) determine if those who participate in a GMI and SOC hand therapy program have differing pain, function, and counts of CRPS diagnoses when compared to those who receive only the SOC. The investigators hypothesize 1) that the project will be feasible to carry out on a larger scale and 2) that an early GMI will improve the pain, functional and upper limb sensorimotor outcomes of persons with closed treatment of DRF relative to a standard of care intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women 55 years or older who have received closed treatment of distal radius fractures

Exclusion Criteria:

* Central nervous system disorders (e.g., Brain injury, Spinal Cord Injury, Parkinson's, Multiple Sclerosis)
* Surgical fixation of fracture
* Non english speaking
* Concomitant ipsilateral injuries (i..e., BBFF)
* Other injuries to the affected limb interfering with baseline affected limb function
* Cognitive disorders which would preclude from following the testing commands and home program participation
* Conditions of the contralateral upper limb which would result in painful and markedly limited active hand, wrist and forearm motion as this may impact the brain's ability to perceive safe and proficient movement during mirror therapy.
* Visual impairments resulting in the inability to participate in GMI components

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in The McGill Pain Scale - Short Form(SF-MPQ) Scores | Change from baseline to 18 weeks
Change in Patient Rated Wrist Evaluation (PRWE) Scores | Change from baseline to 18 weeks
Assessment of Veldman CRPS Type I Diagnostic Criteria | 18 weeks

SECONDARY OUTCOMES:
Change in joint position sense goniometry of wrist and forearm | Change from baseline to 18 weeks
Change in Goniometry of wrist and forearm | Change from baseline to 18 weeks
Change in Grip Dynamometry (% of Unaffected) | Change from baseline to 18 weeks
Therapy Adherence Log | up to 18 weeks
Change in Circumferential Edema measurements of 2nd and 3rd digits | Change from baseline to 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Corey W McGee, PhD, Principal Investigator — University of Minnesota, Program in Occupational Therapy
Locations (1):
- University of Minnesota Program in Occupational Therapy, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Veldman PH, Reynen HM, Arntz IE, Goris RJ. Signs and symptoms of reflex sympathetic dystrophy: prospective study of 829 patients. Lancet. 1993 Oct 23;342(8878):1012-6. doi: 10.1016/0140-6736(93)92877-v. PMID 8105263
- [Background] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870
- [Background] Moseley GL. Graded motor imagery is effective for long-standing complex regional pain syndrome: a randomised controlled trial. Pain. 2004 Mar;108(1-2):192-8. doi: 10.1016/j.pain.2004.01.006. PMID 15109523
- [Background] Lagueux E, Charest J, Lefrancois-Caron E, Mauger ME, Mercier E, Savard K, Tousignant-Laflamme Y. Modified graded motor imagery for complex regional pain syndrome type 1 of the upper extremity in the acute phase: a patient series. Int J Rehabil Res. 2012 Jun;35(2):138-45. doi: 10.1097/MRR.0b013e3283527d29. PMID 22436440
- [Background] King TI 2nd. Circumferential finger measurements utilizing a torque meter to increase reliability. J Hand Ther. 1993 Jan-Mar;6(1):35-6. doi: 10.1016/s0894-1130(12)80179-7. PMID 8343873
- [Background] Walenkamp MM, de Muinck Keizer RJ, Goslings JC, Vos LM, Rosenwasser MP, Schep NW. The Minimum Clinically Important Difference of the Patient-rated Wrist Evaluation Score for Patients With Distal Radius Fractures. Clin Orthop Relat Res. 2015 Oct;473(10):3235-41. doi: 10.1007/s11999-015-4376-9. Epub 2015 Jun 4. PMID 26040969
- [Background] Frenkel MO, Herzig DS, Gebhard F, Mayer J, Becker C, Einsiedel T. Mental practice maintains range of motion despite forearm immobilization: a pilot study in healthy persons. J Rehabil Med. 2014 Mar;46(3):225-32. doi: 10.2340/16501977-1263. PMID 24519331
- [Background] Karagiannopoulos C, Sitler M, Michlovitz S, Tierney R. A descriptive study on wrist and hand sensori-motor impairment and function following distal radius fracture intervention. J Hand Ther. 2013 Jul-Sep;26(3):204-14; quiz 215. doi: 10.1016/j.jht.2013.03.004. Epub 2013 Apr 28. PMID 23628557
- [Background] MacDermid JC, Turgeon T, Richards RS, Beadle M, Roth JH. Patient rating of wrist pain and disability: a reliable and valid measurement tool. J Orthop Trauma. 1998 Nov-Dec;12(8):577-86. doi: 10.1097/00005131-199811000-00009. PMID 9840793
- [Derived] McGee C, Skye J, Van Heest A. Graded motor imagery for women at risk for developing type I CRPS following closed treatment of distal radius fractures: a randomized comparative effectiveness trial protocol. BMC Musculoskelet Disord. 2018 Jun 26;19(1):202. doi: 10.1186/s12891-018-2115-6. PMID 29940926